CLINICAL TRIAL: NCT00205816
Title: An Open-label, Noncomparative, Multi-center, Emergency Use Protocol Administering Tigecycline for the Treatment of Subjects With Infections Due to Resistant Pathogens.
Brief Title: Study Evaluating Emergency-use Tigecycline in Subjects With Resistant Pathogens.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-310
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Bacterial Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Tigecycline

INTERVENTIONS:
Drug: Tigecycline

SUMMARY:
The purpose of this study is to provide a mechanism for the emergency use of tigecycline in the appropriate clinical situations.

The secondary objective is to evaluate the safety and efficacy of tigecycline in the treatment of patients with selected serious infections where other treatment has not been successful.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, greater than 8 years of age and a weight of more than 35 kilograms.
* Patients with current bacterial infections who have not responded to other available appropriate antibiotic therapies.
* Patient must give informed consent.

Exclusion Criteria:

* Patients with an expected survival of less than 2 weeks.
* Patients who have been designated as "Do Not Resuscitate".
* Known or suspected hypersensitivity to tigecycline, tetracyclines, or other compounds related to this class of antibacterial agents.
* Pregnant women or nursing mothers.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
response

SECONDARY OUTCOMES:
micro response at subject level
micro response at pathogen level
clinical response at pathogen level
development of decreased susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- Heidelberg, Germany
- Poland (2):
  - Gdansk
  - Poznan

REFERENCES:
- [Derived] Wallace RJ Jr, Dukart G, Brown-Elliott BA, Griffith DE, Scerpella EG, Marshall B. Clinical experience in 52 patients with tigecycline-containing regimens for salvage treatment of Mycobacterium abscessus and Mycobacterium chelonae infections. J Antimicrob Chemother. 2014 Jul;69(7):1945-53. doi: 10.1093/jac/dku062. Epub 2014 Mar 14. PMID 24633206